CLINICAL TRIAL: NCT02338076
Title: A Study to Document the Effect of Petrolatum on Innate Immune Responses in the Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rockefeller University (Other)
Responsible Party: Principal Investigator, Saakshi Khattri, Sub-investigator, Rockefeller University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EGU-811
Record Dates: First submitted 2015-01-09; First posted 2015-01-14 (Estimated); Results first posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-04

CONDITIONS: Skin Disease
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Interventional arm (Experimental): petrolatum application under occlusion
  Interventions: Drug: Petrolatum application under occlusion

INTERVENTIONS:
Drug: Petrolatum application under occlusion — Day 0 study patients will have 1 patch applied to either back or thighs ( containing 2 wells)
  1 well will be empty and the other well will contain petrolatum
  Day 3 patches will be removed and 3 skin biopsies will be performed 1 biopsy from normal skin at a distance from the patch
  1 biopsy each from under the 2 wells of the patch ( so 1 biopsy from skin that was occluded with petrolatum and 1 biopsy from skin that was occluded without petrolatum)
  Other Names: vaseline under occlusion

SUMMARY:
Petrolatum is a very well-known emollient that has been used since the 1800's. Not only has it been used to help with dry skin, but it is also marketed as a substance that protects minor cuts and burns. In the past it was thought to be inferior to topical antibiotics in infection prevention for cutaneous wounds. However, in 1996 a large, multicenter trial including over 900 patients showed that petrolatum is as safe and effective as the topical antibiotic, bacitracin in preventing infections for patients undergoing dermatological surgery. In this trial, not only did the petrolatum group have similarly low rates of infection, this group also reported no cases of contact dermatitis. Aside from being more expensive than petrolatum, bacitracin and other topical antimicrobials (i.e. neomycin) have been known as common culprits of contact dermatitis. In a study done by the North American Contact Dermatitis Group between 2005-2006, 9.2 and 10% of the over 4,000 patients who were patch tested had an allergic reaction to either bacitracin or neomycin, respectively. For the above reasons, it is clear that petrolatum is an appealing alternative to topical antibiotics for infection prevention in patients undergoing dermatological procedures. This study however lacked any mechanistic analyses to provide molecular insight as to how petrolatum was effective at infection prevention.

The aim of this research is to study the effect of petrolatum on innate immune reactions in the skin. In particular, petrolatum's effect on various antimicrobial peptides after contact with the skin for 3 days will be examined. This will be done through immunohistochemistry for various cellular infiltrates as well as mRNA gene expression via RT-PCR analysis for inflammatory and AMP genes. Tissue samples of petrolatum occluded skin will be compared to both healthy skin and skin under occlusion alone as controls. These comparisons will isolate the effect of the petrolatum on the skin.

DETAILED DESCRIPTION:
Petrolatum (also commonly called Vaseline) is a very well known moisturizer that has been used since the 1800's. Not only has it been used to help with dry skin, but it is also marketed as a substance that protects minor cuts and burns. It is widely used by Dermatologists as a substance to apply to wounds from cutaneous surgical procedures. In a large study, petrolatum was shown to be as effective as one of the major topical antibiotics to help prevent infection in patients who underwent dermatologic procedures. Not only are the other topical antibiotics expensive, but also they are commonly the cause of an allergic reaction in up to 10% of the population. Until now, no reason has been found to explain why petrolatum is effective in infection prevention. In a recent study, skin biopsies of skin that had petrolatum applied to them were obtained. Upon analysis certain "antimicrobial peptides" (peptides that possess anti-bacterial properties that help fight infection) have been found to be elevated. This could provide an answer as to why petrolatum was as effective as the topical antibiotic in the study mentioned above.

This study hopes to improve our understanding of how the immune system acts and how the skin responds to petrolatum. In order to reach this goal, normal volunteers, will be patch tested with petrolatum. Then, biopsies will be taken of the skin at the sites where petrolatum was. Also, small biopsies will be taken from an area that received a patch but no petrolatum and an area that did not receive a patch to serve as controls. The biopsied skin samples will then be studied in a laboratory by methods such as immunohistochemistry and RT-PCR analysis, which will help define the response of the immune system to petrolatum. The rationale for the study is to better define petrolatum's effects in skin and how it is effective at preventing infections.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female between 18 and 85 years of age
* Able to give verbal and written informed consent

Exclusion Criteria:

* Subjects taking any of the following systemic or topical therapies (on the back) within 2 weeks of enrollment: corticosteroids, immunosuppressants, and/or any other medications that may affect the outcome of the study
* subjects with history of keloids
* subjects with self reported history of hepatitis B or C
* HIV positive

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emma Guttman, MD, PhD, Principal Investigator — Rockefeller University
Locations (1):
- The Rockefeller University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Interventional Arm: petrolatum application under occlusion
  Petrolatum application under occlusion: Day 0 study patients will have 1 patch applied to either back or thighs ( containing 2 wells)
  1 well will be empty and the other well will contain petrolatum
  Day 3 patches will be removed and 3 skin biopsies will be performed 1 biopsy from normal skin at a distance from the patch
  1 biopsy each from under the 2 wells of the patch ( so 1 biopsy from skin that was occluded with petrolatum and 1 biopsy from skin that was occluded without petrolatum)
Period: Overall Study
Arm/Group | Interventional Arm
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Interventional Arm
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Expression Levels of Antimicrobial Peptides in Samples of Normal Appearing Skin and Skin Subjected to Occlusion With and Without Petrolatum.
Description: The levels of expression of antimicrobial peptides (S100A8, S100A9, CCL20, PI3, lipocalin , human β-defensin 2 will be measured in skin biopsy samples with petrolatum occlusion, normal skin and occlusion without petrolatum to see if there is any difference in expression Please note- There is only 1 arm with 3 measures - for example, subject 1 had 3 biopsies and the outcome measure S100A8, S100A9, PI3, LIPOCALCIN, HUMAN B DEFENSIN were tested in all 3 biopsies. This is reported as the log of the number of copies. HUMAN B DEFENSIN and CCL20 was not collected. S100A7 and S100A12 were added to the analysis.
Time Frame: 3 days
Measure: Mean (95% Confidence Interval); unit: log of copy number
Groups:
- Interventional Arm With Petrolatum; Arm With Occlusion Only (Without Petrolatum); Control Arm/Normal Skin: petrolatum application under occlusion
  Petrolatum application under occlusion: Day 0 study patients will have 1 patch applied to either back or thighs ( containing 2 wells)
  1 well will be empty and the other well will contain petrolatum
  Day 3 patches will be removed and 3 skin biopsies will be performed 1 biopsy from normal skin at a distance from the patch
  1 biopsy each from under the 2 wells of the patch ( so 1 biopsy from skin that was occluded with petrolatum and 1 biopsy from skin that was occluded without petrolatum)
Arm/Group | Interventional Arm With Petrolatum | Arm With Occlusion Only (Without Petrolatum) | Control Arm/Normal Skin
Number analyzed (Participants) | 20 | 20 | 20
log of copy number
  S100A8 | 9.12 [8.430 to 9.811] | 7.025 [6.334 to 7.716] | 5.415 [4.724 to 6.106]
  S100A9 | 8.926 [8.275 to 9.576] | 6.781 [6.130 to 7.432] | 5.43 [4.779 to 6.081]
  S100A7 | 9.889 [9.500 to 10.476] | 8.883 [8.395 to 9.371] | 8.468 [7.959 to 8.977]
  LIPOCALIN | 10.977 [10.365 to 11.590] | 9.528 [8.916 to 10.141] | 8.182 [7.570 to 8.794]
  S100A12 | 8.795 [8.160 to 9.434] | 8.078 [7.424 to 8.732] | 7.586 [6.814 to 8.358]
  PI3 | 10.555 [10.070 to 11.040] | 8.752 [8.267 to 9.237] | 6.61 [6.126 to 7.095]

2. Primary Outcome: Measurement of Innate Immune Genes (IL6, IL8, and IL1B) in Skin Biopsy Samples With Petrolatum Occlusion, Normal Skin and Occlusion Without Petrolatum to See if There is Any Difference in Expression
Time Frame: 3 days
Measure: Mean (95% Confidence Interval); unit: log of copy number
Arm/Group | Interventional Arm With Petrolatum | Arm With Occlusion Only (Without Petrolatum) | Control Arm/Normal Skin
Number analyzed (Participants) | 20 | 20 | 20
log of copy number
  IL-6 | 10.302 [9.681 to 10.921] | 9.405 [8.790 to 10.019] | 9.100 [8.450 to 9.749]
  IL-8 | 8.205 [7.569 to 8.841] | 6.752 [6.125 to 7.379] | 6.034 [5.413 to 6.655]
  IL-1B | 8.920 [8.284 to 9.583] | 8.145 [7.454 to 8.836] | 7.555 [6.854 to 8.236]

3. Secondary Outcome: Skin Thickness Difference Between Occluded Versus Occluded With Petrolatum Compared With Normal Skin.
Description: skin thickness difference between occluded skin biopsy versus occluded with petrolatum skin biopsy compared with normal skin biopsy was examined
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | Interventional Arm With Petrolatum | Arm With Occlusion Only (Without Petrolatum) | Control Arm/Normal Skin
Number analyzed (Participants) | 20 | 20 | 20
micrometer | 41 (12) | 32 (9) | 24 (8)

4. Secondary Outcome: T-cell Infiltrate in Occluded Versus Occluded With Petrolatum Compared With Normal Skin.
Description: t-cell infiltrate in occluded skin versus occluded with petrolatum skin compared with normal skin ( healthy/not occluded skin)
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: cells per micrometer squared
Arm/Group | Interventional Arm With Petrolatum | Arm With Occlusion Only (Without Petrolatum) | Control Arm/Normal Skin
Number analyzed (Participants) | 20 | 20 | 20
cells per micrometer squared | 1.8421 (4.1801) | 4.5263 (15.6679) | 0.5789 (0.6924)

ADVERSE EVENTS:
Arm/Group | Interventional Arm
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No